CLINICAL TRIAL: NCT01004627
Title: A Prospective Randomized Controlled Trial of the Clinical Effectiveness of Obligatory Versus Elective Duplex Ultrasound Scanning Prior to Arteriovenous Fistula Formation for Haemodialysis Vascular Access in a University Teaching Hospital.
Brief Title: A Study of Routine Versus Selective Use of Ultrasound Scanning Prior to Haemodialysis Fistula Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Access 1
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: End Stage Renal Failure; Surgery
Keywords: fistula; ultrasound; angioaccess; preoperative vein mapping; Haemodialysis; Angioaccess surgery
MeSH Terms: conditions — Renal Insufficiency, Chronic; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group - selective duplex (No Intervention): Patients will receive a duplex ultrasound only if specifically requested following physical examination.
- Obligatory Duplex scan (Experimental): Patients will receive a duplex ultrasound regardless of clinical findings. Arterial and venous duplex ultrasound examination
  Interventions: Procedure: Arterial and venous duplex ultrasound examination

INTERVENTIONS:
Procedure: Arterial and venous duplex ultrasound examination — Ultrasound mapping of all blood vessels in the upper limb of interest
  Arms: Obligatory Duplex scan

SUMMARY:
Dialysis patients have their blood filtered by a machine as their kidneys no longer work. To get blood in and out of these patients it is possible to perform a surgical procedure to increase to size and durability of a vein in the arm to allow repeated needle insertion. This enlarged vein is called a fistula. There is some evidence that ultrasound scanning the blood vessels in the arm before surgery can improve the chances of a successful procedure. The investigators aim to test whether scanning all patients is better than scanning only those who are difficult to assess by physical examination alone.

DETAILED DESCRIPTION:
We will recruit all patients undergoing primary vascular access procedures in our unit who meet inclusion criteria. They will be randomised to either surgery based on clinical findings with duplex ultrasound only if requested by surgeon, or routine duplex ultrasound prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Specific inclusion criteria necessary for invitation to study participation; Patients referred to vascular consultants for primary AV fistula formation (or primary fistula in that limb) for haemodialysis access.

General inclusion criteria;

* Ability to give informed written consent

Exclusion Criteria:

* Specific exclusion criteria;

  * Previous arterial or venous surgery/intervention performed on target limb.
  * Known thrombophilic or thrombotic pathology.
  * Aged under 18 at time of referral

General exclusion criteria;

* Inability to give informed written consent
* Inability to attend follow up appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Primary failure of access (immediate/early thrombosis or failure to mature). | 30 days

SECONDARY OUTCOMES:
Assisted primary patency - being the interval from placement until the time of measurement of patency, including intervening manipulations | open ended
Secondary patency - The interval from placement until time of patency measurement including intervening manipulations | open ended
Site of fistula created | within 1 month of recruitment
Functional primary patency - being the interval from the time of access placement until any intervention designed to maintain or re-establish patency or the time of measurement of patency during which the AVF provides dialysis access. | open ended
Surgeon grade | open ended

OTHER OUTCOMES:
Microparticle concentration | open
  Blood tests will be taken at baseline, 1, 3 and 6 months to investigate the impact of concentrations on patency
Circulating tissue factor concentration | open
  Blood test to be taken at baseline, 1, 3 and 6 months and examined using ELISA to establish the impact of tissue factor concentrations on patency

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Chetter, MBChB FRCS MD, Principal Investigator — Hull University
Locations (1):
- Hull Royal Infirmary, Hull, United Kingdom

REFERENCES:
- [Result] Smith GE, Barnes R, Chetter IC. Randomized clinical trial of selective versus routine preoperative duplex ultrasound imaging before arteriovenous fistula surgery. Br J Surg. 2014 Apr;101(5):469-74. doi: 10.1002/bjs.9435. Epub 2014 Feb 20. PMID 24756913